CLINICAL TRIAL: NCT06015828
Title: Effect of Enteral Bovine Lactoferrin on Neurobehavioral Performance of Preterm Infants
Brief Title: Effect of Enteral Bovine Lactoferrin in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, assistant professor of pediatrics, Ian shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AinShamsUlactoferrin
Record Dates: First submitted 2023-07-16; First posted 2023-08-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded randomized controlled trial Neonates will be randomized using closed envelopes into two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lactoferrin group (Experimental): Neonates will receive a daily dose of 150 mg/kg body weight per day (up to a maximum of 300 mg/day) of bovine lactoferrin and will be prepared for administration by addition by syringe of sterile water (4 mL) orally or through gavage feeding, once the infant's enteral feed volume is more than 12 mL/kg per day until 36 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer. (Asztalos.,et al 2020)
  Interventions: Dietary Supplement: bovine lactoferrin
- control group (No Intervention): Neonates will receive their routine feds and will not receive lactoferrin.

INTERVENTIONS:
Dietary Supplement: bovine lactoferrin — Neonates will receive a daily dose of 150 mg/kg body weight per day (up to a maximum of 300 mg/day) of bovine lactoferrin and will be prepared for administration by addition by syringe of sterile water (4 mL) orally or through gavage feeding, once the infant's enteral feed volume is more than 12 mL/kg per day until 36 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer.
  Arms: lactoferrin group

SUMMARY:
There is a preference for using enteral bovine lactoferrin for preterm infants. Lactoferrin is a sialic acid-rich, iron-binding milk glycoprotein, known to have multifunctional health beneﬁts, including its ability to modulate immune function and facilitate iron absorption, as well as its antibacterial and anti inﬂammatory actions.

The study is an evaluation of the efficacy of enteral bovine lactoferrin on neurobehavioral performance in preterm infants.

DETAILED DESCRIPTION:
Over 15 million infants are born preterm < 37 weeks gestation worldwide. Lactoferrin is about 80- kilo dalton kDa glycoprotein composed of 703 amino acid residues and is a member of the transferrin family, As a member of the transferrin family of iron-binding proteins, lactoferrin shares more than 60% homology at the amino acid level with transferrin and a 77% homology exists between human and bovine species.

Human lactoferrin is the most abundant glycoprotein. It contains 1- 4 Sialic acid residues at the terminal position of N-linked glycan chains for each lactoferrin molecule.

Poly Sialic acid plays a critical role in neural development by modulating the adhesive property of neural cell adhesion molecule and is, therefore, implicated in a wide range of morphogenic events, including cell migration, neuronal outgrowth, path-ﬁnding, sprouting, regeneration, synaptic plasticity, and serving a "reservoir function" for neurotrophic factors. Sia, a key monomeric building block of poly Sialic acid, plays crucial roles in cell-to-cell interactions, neuronal outgrowth, modifying synaptic connectivity, and memory formation An important functional property of lactoferrin is its high afﬁnity for binding iron Iron is a ubiquitous metal that is essential for the function of all mammalian cells. Iron deﬁciency affects neuronal metabolism, neurotransmitter function, and myelination, which have the greatest impact on the brain during early neurodevelopment Lactoferrin is unique in that it contains 2 nutritional molecules of iron and Sialic acid, which are key components involved in early neurodevelopmental and cognitive function for infants Lactoferrin is a bifidogenic glycoprotein found in all vertebrates and mammalian milk, leukocytes, and exocrine secretions Inﬂammation has an adverse impact on cognition, and IL-1β, IL-6, and tumor necrosis factor alpha TNF-α are closely associated with long-term potentiation (LTP) and synaptic plasticity Lactoferrin is an antimicrobial, antioxidant, anti-inflammatory iron-carrying

ELIGIBILITY:
Inclusion Criteria:

* Stable preterm neonates
* gestational age less than 35 weeks
* younger than 72 hours at randomization
* have initiated enteral feds.

Exclusion Criteria:

* 1. Neonates with underlying gastrointestinal problems that prevent oral intake. 2. Neonates with predisposing conditions that profoundly affect growth and development (chromosomal abnormalities,
* structural brain anomalies,
* severe congenital abnormalities). 3. Neonates with a history of perinatal hypoxia. 4. Neonates with a family background of cow milk allergy. 5. Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake.

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
neurobehavioral outcome | at 36 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer.
  The present study is designed to evaluate the effect of oral administration of bovine lactoferrin on the neurobehavioral performance of preterm neonates at 36 weeks corrected age using the Neonatal Intensive Care Unit Neurobehavioral Scale (NNNS). ( minimum 0 , maximum 3 in each category)
Morbidity | At 36 weeks corrected gestational age
  Define any morbidities from oral lactoferrn administration
Mortality | 36 corrected gestational age
  To assess number of deaths in the study group

SECONDARY OUTCOMES:
effect on morbidity and mortality | at 36 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer.
  effect on mortality and major morbidity at 36 weeks corrected gestational age defined as periventricular leukomalacia, necrotizing enterocolitis, and late-onset sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: maha mohamed, PHD, Study Director — Ain Shams University; dina shinkar, PHD, Study Director — Ain Shams University; mariam ibrahim, PHD, Study Director — Ain Shams University; mahmoud kofory, MB.,B.CH, Principal Investigator — Al-Azhar University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt